CLINICAL TRIAL: NCT05621824
Title: A Cohort Study on Screening and Follow-up of High-risk Population of Pancreatic Cancer Based on Endoscopic Ultrasonography
Brief Title: A Cohort Study on Screening and Follow-up of High-risk Population of PDAC Based on EUS
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Tongji Hospital (Other); The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Wu Xi, associate professor, Peking Union Medical College Hospital
Other Study IDs: K2341
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: Early Pancreatic Ductal Adenocarcinoma; Endoscopic Ultrasound; HighRisks for Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal | interventions — Endosonography; Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Baseline sample includes 20ml blood sample, 1 dental plaque sample and 1 stool sample. Follow-up samples include 10mL blood sample, duodenal fluid samples collected during EUS examination and remaining samples of pancreatic puncture tissue and/or cyst fluid during EUS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Solid mass: Patients with solid mass of pancreas during pancreas MR examination.
  Interventions: Device: Endoscopic ultrasound; Procedure: EUS-Fine needle aspiration
- Cystic lesions: Patients with cystic lesions or expansion of MPD during pancreas MR examination.
  Interventions: Device: Endoscopic ultrasound; Procedure: EUS-Fine needle aspiration
- No clear focus: Patients with no clear focus during pancreas MR examination.

INTERVENTIONS:
Device: Endoscopic ultrasound — Use endoscopic ultrasound to examine the pancreatic lesions.
  Groups: Cystic lesions; Solid mass
Procedure: EUS-Fine needle aspiration — If solid mass of pancreas was found during EUS, EUS-FNA shall be conducted for diagnosis.
  Groups: Cystic lesions; Solid mass

SUMMARY:
Study objective: The purpose of this study is to establish a prospective follow-up cohort of high-risk groups of pancreatic cancer, screen early pancreatic cancer through EUS and other means according to the existing clinical process, and evaluate each risk factors. And to prospectively collect biological samples to find molecular markers for early diagnosis of pancreatic cancer.

Study design: This is a real world, multicenter, prospective, observational cohort study.

DETAILED DESCRIPTION:
This study intends to conduct pancreatic MR screening for the high-risk population of pancreatic cancer who meet the requirements and voluntarily participate in this study (see eligibility criteria), and retain baseline information and peripheral blood, dental plaque and stool samples.

I. For patients with solid mass of the pancreas, continue diagnosis and treatment according to the routine clinical path.

II. For patients with MPD dilatation but no clear solid pancreatic mass, EUS examination should be performed after excluding contraindications. During EUS, duodenal fluid samples were collected.

III. If solid mass is found in EUS, FNA shall be performed. If the pathological examination is positive, the patient shall be diagnosed with PDAC and treated according to the clinical routine path of PDAC. If the pathological biopsy sample is negative, repeat FNA after an appropriate interval (1 to 3 months later).

IV. If no solid mass is found in EUS, follow up the patient every 6-12 months for EUS and/or MR examination.

V. For patients with cystic lesions, EUS examination is performed after contraindications are excluded. During EUS, duodenal fluid samples were collected. If solid components such as mural nodules or "worrisome features" are found, FNA will be performed. In order to make a clear diagnosis of some cases, FNA+nCLE will be performed at the same time, and cystic fluid samples will be taken to continue diagnosis and treatment according to the clinical guidelines. If no solid lesions and "worrisome features" are found, follow up the patient every 6-12 months and perform EUS and/or MR examinations.

VI. Follow up and perform pancreatic MR examination every 12 months for those with no clear pancreatic lesions found on pancreatic MR.

The main outcome of this study was the discovery of pancreatic T1 PDAC (tumor diameter < 2cm), or no pancreatic disease was found during the 5-year follow-up period.

The secondary outcome of this study was the discovery of other levels of PDAC, IPMN, chronic pancreatitis, autoimmune pancreatitis and other pancreatic diseases.

The samples involved in this study include baseline and follow-up samples (peripheral blood, dental plaque, stool samples), EUS-FNA solid mass aspiration tissue samples or cystic fluid samples of cystic lesions, and duodenal fluid samples collected during EUS examination. The collected samples were analyzed by transcriptomics, proteomics and next generation sequencing to study the clinical characteristics, molecular, flora markers and gene sequences related to the diagnosis of early pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* From the beginning of the study to the end of the study, the 18-80 year old patients who were admitted to Peking Union Medical College Hospital and related research centers and who met the high-risk population of pancreatic cancer understood and were willing to participate in the study and signed the informed consent form.
* In this study, the high-risk population of pancreatic cancer is defined as patients who meet any of the following conditions:
* A. Patients with previous history of pancreatitis (acute or chronic).
* B. Patients with pancreatic cancer related genetic background, including immediate relatives with a family history of pancreatic cancer. Or genetic syndrome related to pancreatic cancer. [including hereditary breast cancer ovarian cancer syndrome (HBOCS), carney complex (CNC), familial adenomatous polyps (FAP), hereditary diffuse gastric cancer syndrome (HDGC), juvenile polyposis (JPS), cutaneous malignant melanoma (CMM), hereditary papillary renal cell carcinoma (HPRCC) and Lynch syndrome]
* C. Patients with continuous or progressive increase of CA19-9 and CEA.
* D. Patients with potential malignant pancreatic tumors, including mucinous cystic tumor (MCN) and intraductal papillary myxoma of the pancreas (IPMN).
* E. Newly diagnosed patients with diabetes (within 3 years after diagnosis of diabetes).
* F. Other patients who are considered as having high risk factors for pancreatic cancer.

Exclusion Criteria:

* A. Those who are not suitable for endoscopic examination, including but not limited to: poor general condition, serious heart and lung disease, and difficult to tolerate the examination; coagulation disorders; platelets <50 × 10^9/L；those who are not suitable for endoscopic examination after interview by an endoscopic physician.
* B. The patient or family member could not understand the conditions and objectives of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high risks for pancreas cancer in Peking Union Medical College Hospital and other related research centers in China.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with T1 PDAC | 5 years
  Patients found with early stage PDAC, which means tumor size < 2cm.
Number of Participants with no clear pancreas lesions | 5 years
  Patients found with no clear pancreas lesions during 5 years follow-up.

SECONDARY OUTCOMES:
Number of Participants with other stages of PDAC | 5 years
  Patients found with any other stages of PDAC except from T1 PDAC.
Number of Participants with IPMN | 5 years
  Patients found with IPMN during the study.
Number of Participants with chronic pancreatitis | 5 years
  Patients found with chronic pancreatitis during the study.
Number of Participants with autoimmune pancreatitis | 5 years
  Patients found with autoimmune pancreatitis during the study.
Number of Participants with other pancreas diseases | 5 years
  Patients found with any other pancreas diseases except from listed above during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Xi Wu, M.D., Study Director — Peking Union Medical College Hospital; Shengyu Zhang, M.D., Principal Investigator — Peking Union Medical College Hospital; Yuheng Zhang, MD candidate, Principal Investigator — Peking Union Medical College Hospital